CLINICAL TRIAL: NCT02840344
Title: Couples-Based Mindfulness for Young Breast Cancer Survivors
Acronym: C-MBSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Missouri, St. Louis (Other); University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Ann Bettencourt, Dr. Ann Bettencourt, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003808
Record Dates: First submitted 2016-06-29; First posted 2016-07-21 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: Couple Functioning; Stress Reduction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couples MBSR (Experimental): Young breast cancer survivors and their partners take part in an 8-week Couples Mindfulness-Based Stress reduction (C-MBSR) intervention. The course will be taught through recorded videos of a trained MBSR instructor. The young breast cancer survivor and partner will be asked to watch a video module, together, each week for a total of 8 weeks. The C-MBSR course consists of practicing mindful stress reduction techniques and filling out handouts.
  Both members of the couple will be asked to complete surveys assessing primary and secondary outcome measures administered at baseline and after final session. Participants will be asked to provide a Salivary Cortisol sample at baseline and after the 8th session. Follow up Surveys will be administered at one and three months after intervention.
  Interventions: Behavioral: Couples MBSR
- Individual MBSR (Active Comparator): Young breast cancer survivors take part in an 8-week Individual Mindfulness-Based Stress reduction (I-MBSR) intervention. The course will be taught through recorded videos of a trained MBSR instructor. The young breast cancer survivor will be asked to watch a video module each week for 8 weeks in a row. The I-MBSR course consists of practicing mindful stress reduction techniques and filling out handouts.
  Both members of the couple will be asked to complete surveys assessing primary and secondary outcome measures administered at baseline and after final session. Participants will be asked to provide a Salivary Cortisol sample at baseline and after the 8th session. Follow up Surveys will be administered at one and three months after intervention.
  Interventions: Behavioral: Individual MBSR

INTERVENTIONS:
Behavioral: Couples MBSR — Both members of the couple will be asked to participate in the weekly video sessions and activities.
  Arms: Couples MBSR
Behavioral: Individual MBSR — Only the young breast cancer survivor will participate in the weekly video sessions and activities.
  Arms: Individual MBSR

SUMMARY:
This study aims to improve relationship, psychological, and physical adjustment among young breast cancer survivors (YBCS; diagnosed at age 45 or younger) and their committed/life partners. A mindfulness-based stress reduction (MBSR) intervention has been designed to meet the specific needs for young breast cancer survivors and their partners. The intervention will be administered in your home by using recorded videos of a trained MBSR instructor. Before, during, and after the 8-week intervention, participants will be asked to complete surveys.

DETAILED DESCRIPTION:
Participants will be young breast cancer survivors (YBCS) and their partners. Young breast cancer survivors are those diagnosed at age 45 or younger. This study includes stress reducing interventions known to have a positive influence on physical and psychological functioning that will be administered through recorded videos. The interventions include watching an hour-long video stress-reduction class, each week, for 8 weeks and practicing guided meditations. YBCS participants will be randomly assigned to either an 8-week mindfulness-based stress reduction course designed for couples (C-MBSR) or an 8-week mindfulness-based stress reduction course for individuals. At the end of the study all participants (regardless of what assignment) will receive both sets of stress-reducing videos. Partners of the YBCS assigned to the couples condition will also be asked to watch the 8 C-MBSR videos. Some young breast cancer survivor participants and their partners will be asked to complete provide salivary cortisol and all survivors and partners will be asked to complete the 4 surveys.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years to 45 years old when diagnosed with breast cancer
2. Diagnosed with stage 0, I, II, III breast cancer
3. within 1 to 6 years after diagnosis of breast cancer
4. Married or unmarried and living together.
5. Living anywhere in the United States
6. Both members of the couple must understand, read, and speak English
7. Both members of the couple must have regular access to email and willingness to use the Internet.

Exclusion Criteria:

1. Neither members of the couple may be experienced meditators (20 minutes daily, 5 days a week or more, for over a year) or graduates of a former MBSR class.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Change in couple functioning measured by the Measured by the Dyadic Adjustment Scale | Baseline to 6 months
  The scale scores will be the average of items in the measure. The scale scores will be averaged to create a summary score for each condition (no individual scores will be reported).
Change in couple functioning measured by the Measured by the Autonomy and Relatedness Inventory | Baseline to 6 months
  The scale scores will be the average of items in the measure. The scale scores will be averaged to create a summary score for each condition (no individual scores will be reported).
Change in couple functioning measured by the Sexual Interest and Satisfaction Scale | Baseline to 6 months
  The scale scores will be the average of items in the measure. The scale scores will be averaged to create a summary score for each condition (no individual scores will be reported).
Change in couple functioning measured by the Interpersonal Mindfulness Scale | Baseline to 6 months
  The scale scores will be the average of items in the measure. The scale scores will be averaged to create a summary score for each condition (no individual scores will be reported).
Perceived Partner Responsiveness | Baseline to 8 weeks
  This scale will be measured each week for the 8 weeks of the intervention

SECONDARY OUTCOMES:
Change in anxiety scores measured by PROMIS -- Anxiety | Baseline to 6 months
  The scale scores will be the average of items in the measure. The scale scores will be averaged to create a summary score for each condition (no individual scores will be reported).
Change in depression scores measured by the PROMIS -- Depression | Baseline to 6 months
  The scale scores will be the average of items in the measure. The scale scores will be averaged to create a summary score for each condition (no individual scores will be reported).
Change in fatigue scores measured by PROMIS -- Fatigue | Baseline to 6 months
  The scale scores will be the average of items in the measure. The scale scores will be averaged to create a summary score for each condition (no individual scores will be reported).
Change in stress scores measured by the Perceived Stress Scale | Baseline to 6 months
  The scale scores will be the average of items in the measure. The scale scores will be averaged to create a summary score for each condition (no individual scores will be reported).
Changes in physical functioning measured by the PROMIS - Physical Function | Baseline to 6 months
  The scale scores will be the average of items in the measure. The scale scores will be averaged to create a summary score for each condition (no individual scores will be reported).
Changes in salivary cortisol biomarker to assess stress levels | Baseline to 8 weeks
  Saliva will be analyzed for cortisol and summary scores will be calculated for each condition (no individual scores will be reported).
Changes in trait mindfulness measured by Mindful Attention and Awareness Scale | Baseline to 6 months
  The scale scores will be the average of items in the measure. The scale scores will be averaged to create a summary score for each condition (no individual scores will be reported).

CONTACTS AND LOCATIONS:
Overall Officials: Ann Bettencourt, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No